CLINICAL TRIAL: NCT02440334
Title: Two and Three Dimensional Contrast-Enhanced Ultrasound for Screening of Renal Cell Carcinoma Recurrence Following Cryoablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, john eisenbrey, Research Assistant Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15P.039; JT 7277 (Other: JeffTrial Number)
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma
Keywords: cryosurgery; ultrasonography
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Contrast Ultrasound Reccurence Screening (Experimental): Patients scheduled for MRI/CT follow up of a renal cancer previously treated by cryoablation therapy who will also undergo a contrast-enhanced ultrasound exam. This is a one-time imaging study and contrast ultrasound exams will be compared to the clinically scheduled MRI/CT.
  Interventions: Drug: Optison

INTERVENTIONS:
Drug: Optison — Optison is an ultrasound contrast agent. The agent is a blood pooling agent administered via catheter and provides improved ultrasound visualization of the vasculature.

SUMMARY:
The purpose of the proposed trial is to determine whether contrast-enhanced ultrasound (CEUS) can be used to assess the recurrence of renal cell carcinoma (RCC) after cryoablation compared to contrast enhanced CT or MR (the standard evaluation). This study involves the off-label use of an FDA-approved ultrasound contrast agent, Optison that flows in the vascularity. CEUS will be performed by both two and three dimensional ultrasound to examine post-cryoablation vascularity changes to screen for recurrent disease.

DETAILED DESCRIPTION:
Subjects eligible for trial enrollment will be identified by the Thomas Jefferson University Urology group from their patient population of subjects under active surveillance for recurrence of a previously cryoablated RCC. A research coordinator will explain the study to the patient. The patient will be given time to consider the risks and benefits of the study and ask questions about participation. The coordinator will review the consent form with the patient and then the patient will be given the form to review. The patient, coordinator, and a study investigator will all sign the consent form. The patient will be given a copy of the signed consent form for their records.

Screening assessments will be performed prior to CEUS imaging. Trial participants will have the presence of inclusion criteria and absence of exclusion criteria verified by providing a medical history. A full demographic profile, known drug allergies or intolerances, and a review of the subject's medical/surgical history will be recorded. If the subject is a woman of childbearing age, she will have a urine pregnancy test (the results of which will be made available to the subject prior to study initiation).

All contrast injections will be supervised by a board certified physician. Resuscitation equipment and trained personnel will be in immediate proximity to the patient during each CEUS exam. The ultrasound examinations will be performed by a qualified sonographer. Ultrasound exams will take place the morning prior to the patient's 8, 12, 18, 24, or 36 month CT/MRI follow up (scheduled as part of their clinical care) or during their consultation in Jefferson's Urology clinic (for patients who have imaging performed outside Jefferson). Procedures and equipment for this trial will be used in accordance with typical clinical procedures. All trial procedures will be conducted in accordance with Good Clinical Practice. For the ultrasound examination, the patient will be asked to lie in the supine position and a catheter will be placed in a superficial vein (preferably an antecubital vein). Acoustic coupling gel will be applied to the area of interest. A state of the art ultrasound scanner with 2D and 3D curvilinear probes will be used.

A baseline ultrasound grayscale scan will be used to identify the tumor and to evaluate the following criteria: size, shape, and orientation of the lesion; echogenicity compared to surrounding tissue. Standard power Doppler of the lesion will also be performed. When possible, previous MR/CT data will be uploaded onto the scanner in order to perform image fusion for ultrasound guidance during imaging. The distribution of color signals and the overall color content of the tumor will be evaluated by comparing the pattern and amount of color to the normal surrounding tissue. Following baseline scanning, patients will receive a 1 ml intravenous injection of Optison (GE Healthcare, Princeton, NJ) in a peripheral vein followed by renal mass imaging in 2D CHI (a nonlinear contrast imaging package). Ten minutes after the 2D CEUS exam, patients will receive a second bolus injection of Optison followed by 3D CHI (using a curvilinear 3D array). All contrast injections will be supervised by a board certified physician. Resuscitation equipment and trained personnel will be immediate proximity to the patient during each contrast-enhanced ultrasound exam. Digital clips of the exams will be recorded through the contrast agent wash-in and wash-out phases for at least two minutes and stored for later use. The subject will then be monitored for adverse reactions for 30 minutes. If the patient wishes to continue participating in the study, they will be eligible for CEUS exams during their future clinically scheduled follow up exams as long as these take place within the study timeframe.

Patients will be monitored for AEs during and 30 minutes after contrast administration. All other procedures will be performed according to standard of care. No further patient monitoring is required as side effects of Optison are acute in nature and no renal toxicity has been reported.

ELIGIBILITY:
Inclusion Criteria:

* Previously received cryotherapy of RCC.
* Be scheduled for contrast-enhanced MRI/CT to monitoring of RCC recurrence as part of their 8, 12, 18, 24, or 36 month CT/MRI follow up.
* Be at least 18 years of age.
* Be medically stable.
* If a female of child-bearing age, must have a negative pregnancy test.
* Have signed Informed Consent to participate in the study.

Exclusion Criteria:

* Females who are pregnant or nursing.
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
* Patients on life support or in a critical care unit.
* Patients with unstable occlusive disease (eg, crescendo angina)
* Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia.
* Patients with uncontrolled congestive heart failure (NYHA Class IV)
* Patients with recent cerebral hemorrhage.
* Patients with known sensitivities to albumin, blood, or blood products
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination.
* Patients with known hypersensitivity to perflutren
* Patients with cardiac shunts.
* Patients with congenital heart defects.
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli.
* Patients with respiratory distress syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Eisenbrey JR, Shaw CM, Lyshchik A, Machado P, Lallas CD, Trabulsi EJ, Merton DA, Fox TB, Liu JB, Brown DB, Forsberg F. Contrast-Enhanced Subharmonic and Harmonic Ultrasound of Renal Masses Undergoing Percutaneous Cryoablation. Acad Radiol. 2015 Jul;22(7):820-6. doi: 10.1016/j.acra.2015.03.008. Epub 2015 Apr 14. PMID 25882093

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contrast Ultrasound Reccurence Screening
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Contrast Ultrasound Reccurence Screening
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: The Sensitivity of Detecting RCC Recurrence (Using Contrast-enhanced MRI as a Reference Standard) on a Single Contrast-enhanced Ultrasound Exam.
Description: Patients scheduled for follow up contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) of a previously cryoablatated renal cell carcinoma (RCC) through Thomas Jefferson University's Urology clinic will undergo a single ultrasound exam using contrast enhanced ultrasound. Ultrasound imaging will be performed using a state of the art ultrasound scanner with two and three dimensional curvilinear transducers.
Time Frame: 8 months post cryoblation
Measure: Number; unit: percent of patients
Arm/Group | Contrast Ultrasound Reccurence Screening
Number analyzed (Participants) | 53
percent of patients | 100

ADVERSE EVENTS:
Time Frame: Each participant was monitored for 30 minutes following Optison Injection.
Arm/Group | Contrast Ultrasound Reccurence Screening
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT02440334/Prot_SAP_000.pdf